CLINICAL TRIAL: NCT04935450
Title: Pulmonary Inflammation Profiles in COVID-19 Related ARDS
Brief Title: Pulmonary Inflammation in COVID-19 ARDS
Acronym: IMPU-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Tommaso Bardi, Principal Investigator, Hospital Universitario Ramon y Cajal
Other Study IDs: 398-20
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: ARDS Due to Disease Caused by Severe Acute Respiratory Syndrome Coronavirus 2; COVID-19 Acute Respiratory Distress Syndrome
Keywords: ARDS; COVID-19; Broncho Alveolar Lavage; Pulmonary Inflammation; Mechanical Ventilation; Respiratory Mechanics
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalveolar Lavage Fluid samples Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bronchoalveolar lavage — Low volume Broncho alveolar lavage. During optic flexible bronchoscopy through the tracheal tube or the tracheostomy cannula a maximum of 4 aliquots of 20 ml normal saline will be instilled in a wedged position in the right medium lobe of the patients and then aspirated untill reaching a total of 25ml of fluid (BALF) for analysis

SUMMARY:
Patients older than 18 years of age, with COVID-19 related ARDS (C-ARDS) hospitalized in the ICU and invasively mechanically ventilated will be included in the study.

This is an observational cohort study. After informed consent by the next of kin, and within the first 72 hours of invasive mechanical ventilation a blood and a Broncho Alveolar Lavage Fluid (BALF) sample will be collected. If the patients remain invasively mechanically ventilated a second and third blood and BALF sample will be collected every 7-10 days.

DETAILED DESCRIPTION:
The main objective of the core study is to measure a number of biochemical, cellular and inflammatory mediators in the BALF of C-ARDS patients and evaluate their correlation with the course of disease in terms of respiratory mechanics, complications and outcomes.

The mediators selected have been previously used in ARDS investigation to attempt prognostic and predictive enrichment.

Patients hospitalized in the ICU following C-ARDS and requiring invasive mechanical ventilation will be candidates for enrollment.

Patients enrolled in the study (Informed consent obtained from next of kin) will be subject to the realization of optic bronchoscopy within the first 72 h of mechanical ventilation to obtain BALF for analysis. A second and third bronchoscopy and sampling of BALF will be performed every 7-10 days if mechanical ventilation and the clinical conditions allow it. A sample of whole blood will be taken contemporary to each bronchoscopy in order to perform parallel measurements (lungs and peripheral blood). Patients will be followed up until hospital discharge.

BALF samples will be divided to perform different analysis in the immunology, cytology and microbiology labs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* COVID-19 related ARDS
* Hospitalized in ICU
* Invasive mechanical ventilation

Exclusion Criteria:

* Immunocompromised for previous condition
* transplanted patients
* Known pulmonary bacterial co-infection at the time of admission to the ICU
* Contraindication to the realization of Bronchoscopy (Itracranial Hypertension, severe hypoxaemia with P/F < 80, severe hemodynamic instability, severe arrhythmia, non correctable coagulopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 ARDS ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-08-16 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 3 months
  Correlation of BALF and Blood mediators with ICU mortality

SECONDARY OUTCOMES:
Respiratory mechanics | Day 0 (after study inclusion) and every day up to 3 months
  Correlation of BALF and Blood mediators with respiratory mechanics during invasive mechanical ventilation
BALF PCR | Day 0 (performance of first BALF sample) Day 8, Day 16
  Semiquant PCR of SARS-CoV-2 in bronchoalveolar lavage fluid, comparison with contemporary PCR in Blood
BALF characteristics | Day 0 (performance of first BALF sample) Day 8, Day 16
  Cellular populations in BALF and their change over time
BALF cytoquines | Day 0 (performance of first BALF sample) Day 8, Day 16
  Cytoquines in BALF and change over time

OTHER OUTCOMES:
Hospital Mortality | Up to 3 months
  Mortality in hospital
Health related quality of life via SF-36 questionnaire | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No